CLINICAL TRIAL: NCT03402854
Title: tDCS and Bimanual Therapy for Children With Hemiplegic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Collaborators: University of Minnesota (Other); Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS_bimanual
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy; Spastic Hemiplegic Cerebral Palsy; Spastic Hemiparesis; Spastic Hemiplegia
Keywords: pediatric; children; non-invasive brain stimulation; transcranial direct current stimulation; bimanual training; hand training
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Children will be randomly allocated to one of two parallel arms of the study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and care providers will not be told of their group allocation. Participants in the sham group will receive a brief stimulation of the scalp, which will give them a feeling of being stimulated. This sham stimulation has been shown to effectively blind participants to group. Assessors will not be told the type of study being conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS + bimanual training (Experimental): In this arm, participants will engage in 120 min of bimanual training. Bimanual training involves using both hands to play with toys and games during the study. During the first 20 min of bimanual training, participants will receive active tDCS via sponges over the scalp.
  Interventions: Device: active transcranial direct current stimulation; Behavioral: bimanual training
- Sham tDCS + bimanual training (Experimental): In this arm, participants will engage in 120 min of bimanual training. Bimanual training involves using both hands to play with toys and games during the study. During the first 20 min of bimanual training, participants will wear the tDCS device that is worn by the active tDCS group, but in the sham group, participants will not receive stimulation during this 20 min period.
  Interventions: Behavioral: bimanual training

INTERVENTIONS:
Device: active transcranial direct current stimulation — Participants will receive 20 min of tDCS over the scalp during the first 20 min of bimanual training.
  Arms: Active tDCS + bimanual training
Behavioral: bimanual training — Participants will engage in movements that use both hands, by playing with toys and games.

SUMMARY:
The goal of this study is to test the efficacy of transcranial direct current stimulation combined with bimanual training on hand function in children with unilateral spastic cerebral palsy (USCP). Children who enroll in the protocol will be randomized to receive either sham (not stimulating) tDCS plus bimanual training, or active (stimulating) tDCS plus bimanual training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital hemiplegic cerebral palsy
* Ability to lift and grasp light objects with affected hand
* Ability to extend wrist of affected hand 15 degrees
* Ability to follow instructions and provide informed assent
* Parent(s) able to provide informed consent

Exclusion Criteria:

* Seizures after age 2 years
* Spasticity medication within 6 months before study
* Selective dorsal rhizotomy
* Surgery in affected upper extremity within year before study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Assisting Hand Assessment | Day before intervention begins, compared to day after intervention ends (six days after intervention begins)
  Measure of how well the child uses both hands cooperatively for bimanual activities

SECONDARY OUTCOMES:
Jebsen-Taylor Test of Hand Function | Day before intervention begins, compared to day after intervention ends (six days after intervention begins)
  Measure of movement speed of affected hand
Box and Blocks test | Day before intervention begins, compared to day after intervention ends (six days after intervention begins)
  Measure of movement speed of affected hand

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Friel, PhD, Principal Investigator — Burke Medical Research Institute
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share IPD via the NIH Data Hub (DASH), which is sponsored by NICHD.
Time Frame: Data will be available when study is complete, and remain in DASH indefinitely.

REFERENCES:
- [Background] Gordon AM, Ferre CL, Robert MT, Chin K, Brandao M, Friel KM. HABIT+tDCS: a study protocol of a randomised controlled trial (RCT) investigating the synergistic efficacy of hand-arm bimanual intensive therapy (HABIT) plus targeted non-invasive brain stimulation to improve upper extremity function in school-age children with unilateral cerebral palsy. BMJ Open. 2022 Feb 21;12(2):e052409. doi: 10.1136/bmjopen-2021-052409. PMID 35190424